CLINICAL TRIAL: NCT05533827
Title: The Effect of Distraction Technique on Children's Pain, Anxiety and Fear of Medical
Brief Title: The Effect of Distraction Technique on Children's Pain, Anxiety and Fear of Medical Procedure in Invasive Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Nursen Goktas, Registered Nurse, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BandirmaOnyediEylulUU
Record Dates: First submitted 2022-08-17; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Child Behavior
Keywords: music; Kaleidoscope; virtual reality glasses
MeSH Terms: conditions — Child Behavior | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Kaleidoscope (Experimental): Kaleidoscope
  Interventions: Other: Kaleidoscope; Other: Music; Other: Virtual reality glasses
- Music (Experimental): Music listening
  Interventions: Other: Kaleidoscope; Other: Music; Other: Virtual reality glasses
- Virtual reality glasses (Experimental): Virtual reality glasses
  Interventions: Other: Kaleidoscope; Other: Music; Other: Virtual reality glasses
- Control (No Intervention): Control

INTERVENTIONS:
Other: Kaleidoscope — Kaleidoscope
  Arms: Kaleidoscope; Music; Virtual reality glasses
Other: Music — Music
  Arms: Kaleidoscope; Music; Virtual reality glasses
Other: Virtual reality glasses — Virtual reality glasses
  Arms: Kaleidoscope; Music; Virtual reality glasses

SUMMARY:
This study was conducted on the effects of visual and/or auditory distraction techniques applied to children aged 7-12 years who applied to Çanakkale Mehmet Akif Ersoy State Hospital Gynecology and Pediatric Emergency Service during invasive procedures (blood sampling, intravenous access or intramuscular injection in the deltoid region). Kaleidoscope, music concert, virtual reality glasses) is a randomized controlled experimental study to determine the effect of children on pain, anxiety and fear of medical procedures.

ELIGIBILITY:
Inclusion Criteria:

* The child is between the ages of 7 and 12
* Admission of the child to the pediatric emergency service for diagnosis and treatment
* The child's general condition is stable
* Deciding on one of the interventions such as blood collection, vascular access, deltoid region intramuscular injection after the examination, and the absence of any other invasive intervention planning
* The fact that the invasive intervention was performed in one go
* The child does not have vision and hearing problems
* The child has no pain (due to the disease, drug side effects, distension)
* The child does not have a chronic disease (kidney, diabetes, etc.) that will require frequent invasive procedures.
* The child's mental development level to be able to answer the questions asked
* The child and parent speak and understand Turkish comfortably
* The children and their parents are willing to participate in the research.
* Parents give written consent

Exclusion Criteria:

* The child has a history of epilepsy, vertigo and neurological disease
* Having a history of fainting during blood draw
* Having a disease that causes chronic pain
* Wearing glasses or hearing aids
* Complication development during invasive intervention (allergy, syncope, etc.)
* If the child is in danger of life and is taken to the very urgent patient examination room (resuscitation room)
* Deciding that the child is a forensic case after the examination

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Pain level | 5 minutes before intervention
  Pain level
Pain level | 5 minutes after intervention
  Pain level
Anxiety level | 5 minutes before intervention
  Anxiety level
Anxiety level | 5 minutes after intervention
  Anxiety level
Fear of medical procedures | 5 minutes before intervention
  Fear of medical procedures
Fear of medical procedures | 5 minutes after intervention
  Fear of medical procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Banıdrma Onyedi Eylul University, Bandırma, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided